CLINICAL TRIAL: NCT00025506
Title: A Phase II Evaluation of Thalidomide (NSC #66847) in the Treatment of Recurrent or Persistent Carcinosarcoma of the Uterus
Brief Title: Thalidomide in Treating Patients With Recurrent or Persistent Carcinosarcoma of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02421; NCI-2012-02421 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068967; GOG-0230B (Other: Gynecologic Oncology Group); GOG-0230B (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Thalidomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Thalidomide — Given orally
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Softenon; Synovir; Talimol; Thalomid

SUMMARY:
This phase II trial is studying how well thalidomide works in treating patients with carcinosarcoma of the uterus that has come back or that does not go to remission (decrease or disappear but may still be in the body) despite treatment. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the antitumor cytostatic activity of thalidomide, as measured by the probability of progression-free survival (PFS) for at least 6 months, in patients with recurrent or persistent uterine carcinosarcoma.

II. Determine the nature and degree of toxicity of this drug in these patients.

Secondary I. Determine the partial and complete response rates in patients treated with this drug.

II. Determine the duration of PFS and overall survival of patients treated with this drug.

III. Determine the effect of this drug on initial performance status and histological grade in these patients.

IV. Correlate serum and plasma biomarkers, including vascular endothelial growth factor and basic fibroblast growth factor, with clinical outcome (i.e., PFS) in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uterine sarcoma

  * Carcinosarcoma (malignant mixed müllerian tumor)

    * Homologous or heterologous type
* Recurrent or persistent with documented disease progression after prior local therapy
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI
  * At least 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are considered non-target lesions
* Must have received 1 prior initial chemotherapy regimen (including high-dose ,consolidation, or extended therapy after surgical or nonsurgical assessment) for carcinosarcoma
* No documented brain metastases since diagnosis of cancer

  * Patients with stable CNS deficits are allowed provided that there is no evidence of brain metastases on CT scan or MRI
* Ineligible for a higher priority Gynecologic Oncology Group (GOG) protocol (if one exists), including any active phase III GOG protocol for the same patient population
* Performance status - GOG 0-2 if received 1 prior therapy regimen
* Performance status - GOG 0-1 if received 2 prior therapy regimens
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance greater than 60 mL/min
* Not pregnant
* Negative pregnancy test
* Fertile patients must use at least 1 highly active method of contraception and 1 additional effective method of contraception for at least 4 weeks before, during, and for at least 4 weeks after study participation
* No seizure disorders since diagnosis of cancer

  * Patients with a history of seizure disorders are allowed provided that the seizures have been stable (i.e., no seizure within the past 12 months) while on an appropriately monitored treatment regimen
* No active infection requiring antibiotics
* No greater than grade 1 sensory or motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 3 weeks since prior immunologic agents for uterine sarcoma
* No prior thalidomide
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for uterine sarcoma and recovered
* No more than 1 prior cytotoxic chemotherapy regimen for recurrent or persistent uterine sarcoma
* No prior non-cytotoxic chemotherapy for recurrent or persistent uterine sarcoma
* No concurrent bisphosphonates (e.g., zoledronate)
* At least 1 week since prior hormonal therapy for uterine sarcoma
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for uterine sarcoma and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas
* See Disease Characteristics
* Recovered from prior surgery
* At least 3 weeks since any other prior therapy for uterine sarcoma
* No prior anticancer therapy that would preclude study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2001-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. McMeekin, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/4/2001 and closed to accrual on 3/3/2008 (suspended from 6/30/2003 to 8/1/2005).
Groups:
- Thalidomide: Thalidomide 200 mg PO once a day initial dose (each 28-day period will be considered one cycle). Dose increased by 200 mg every 2 weeks to maximum dose of 1000 mg/day until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Thalidomide
Started | 55
Completed | 45 (Eligible and treated patients.)
Not Completed | 10
Not completed — Ineligible: clerical error | 1
Not completed — Ineligible: wrong cell type | 5
Not completed — Ineligible: inadequate pathology | 2
Not completed — Never Treated | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.9)
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 1
  50-59 years | 7
  60-69 years | 23
  70-79 years | 11
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
Histologic type [Number; unit: participants]
  Carcinosarcoma-homologous | 22
  Carcinosarcoma-heterologous | 16
  Carcinosarcoma, MMT | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) > 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle for 6 months
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
percentage of participants | 17.8 [9 to 30]

2. Primary Outcome: Frequency and Severity of Adverse Effects as Assessed by Common Toxicity Criteria (CTC) v2.0
Time Frame: Each cycle during treatment and 30 days after the last treatment (average 4 months)
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the adverse event.
- Grade 1: Number of patients who experienced a Grade 1 adverse event (Common Toxicity Criteria version 2)
- Grade 2: Number of patients who experienced a Grade 2 adverse event (Common Toxicity Criteria version 2)
- Grade 3: Number of patients who experienced a Grade 3 adverse event (Common Toxicity Criteria version 2)
- Grade 4: Number of patients who experienced a Grade 4 adverse event (Common Toxicity Criteria version 2)
Arm/Group | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 45
Participants
  Nausea | 31 | 4 | 6 | 4 | 0
  Vomiting | 36 | 4 | 4 | 1 | 0
  Constipation | 27 | 6 | 9 | 3 | 0
  Anorexia | 42 | 2 | 1 | 0 | 0
  Fatigue | 22 | 5 | 15 | 3 | 0
  Neutropenia | 41 | 1 | 3 | 0 | 0
  Thrombocytopenia | 44 | 1 | 0 | 0 | 0
  Anemia | 22 | 9 | 9 | 4 | 1
  Cardiovascular | 31 | 9 | 2 | 1 | 2
  Neuropathy (sensory) | 27 | 12 | 5 | 1 | 0
  Other neurologic | 31 | 2 | 6 | 6 | 0
  Dermatologic | 39 | 4 | 2 | 0 | 0
  Metabolic | 40 | 3 | 0 | 2 | 0
  Pain | 38 | 4 | 2 | 1 | 0

3. Secondary Outcome: Progression Free Survival
Description: as for outcome 1
Time Frame: Every other cycle until progression or death, up to 5 years.
Population: Eligible and treated patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
months | 1.91 [1.35 to 4.17]

4. Secondary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: For those patients whose disease can be evaluated by physical examination, response was assessed prior to each 28-day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle. (average = 4 months)
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
percentage of participants | 4.4 [1 to 13]

5. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
months | 5.9 [3.6 to 9.6]

6. Secondary Outcome: Initial Performance Status
Description: Performance status 0 = Fully active, able to carry on all pre-disease performance without restriction.
  Performance status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work.
  Performance status 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: baseline
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
Participants
  Performance status = 0 | 30
  Performance status = 1 | 12
  Performance status = 2 | 3

7. Secondary Outcome: Initial Histologic Grade
Description: G3 - Predominantly solid or entirely undifferentiated carcinoma. Not graded - tumor grade not reported.
Time Frame: Baseline
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Thalidomide
Number analyzed (Participants) | 45
Participants
  Grade 3 | 4
  Not graded | 41

8. Other Pre Specified Outcome: Serum and Plasma Concentrations of VEGF and bFGF With PFS
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Serum and Plasma Concentrations of Vascular Endothelial Growth Factor (VEGF) and bFGF
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) for up to 5 years after stopping study treatment.
Arm/Group | Thalidomide
Serious Adverse Events (participants affected / at risk) | 15/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide (N=45)
Thrombosis Embolism (Cardiac disorders) | 2
Constitutional Symptoms Other (General disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Gi Other (Gastrointestinal disorders) | 1
Hemorrhage With Grade 3/4 Thrombocytopenia (Vascular disorders) | 1
Bilirubin (Hepatobiliary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide (N=45)
Inner Ear/Hearing (Ear and labyrinth disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Transfusion Prbc's (Blood and lymphatic system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 29
Transfusion Platelets (Blood and lymphatic system disorders) | 1
Arrhythmia Nodal/Junctional Dysrhythmia (Cardiac disorders) | 1
Edema (Cardiac disorders) | 12
Thrombosis Embolism (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Fever(No Neutropenia) (General disorders) | 2
Weight Gain(No Vod) (General disorders) | 1
Constitutional Symptoms Other (General disorders) | 2
Sweating (General disorders) | 1
Fatigue (General disorders) | 24
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash Desquamation (Skin and subcutaneous tissue disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Hot Flashes/Flushes (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Diarrhea With Colostomy (Gastrointestinal disorders) | 1
Mouth Dryness (Gastrointestinal disorders) | 4
Ascites Non-Malignant (Gastrointestinal disorders) | 4
Taste Disturbance (Gastrointestinal disorders) | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 20
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 16
Gi Other (Gastrointestinal disorders) | 5
Rectal Bleeding/Hematochezia (Vascular disorders) | 1
Epistaxis (Vascular disorders) | 1
Vaginal Bleeding (Vascular disorders) | 2
Hematuria No Vaginal Bleeding (Vascular disorders) | 2
Hepatic Other (Hepatobiliary disorders) | 1
Hypoalbuminemia (Hepatobiliary disorders) | 4
Sgot(Ast) (Hepatobiliary disorders) | 1
Alkaline Phosphatase (Hepatobiliary disorders) | 3
Bilirubin (Hepatobiliary disorders) | 2
Infection Without Neutropenia (Infections and infestations) | 3
Lymphatics (Blood and lymphatic system disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolic Other (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesmia (Metabolism and nutrition disorders) | 3
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Hallucinations (Nervous system disorders) | 1
Depressed Level Of Consciousness (Nervous system disorders) | 8
Cognitive Disturbance (Nervous system disorders) | 1
Ataxia(Incoordination) (Nervous system disorders) | 2
Mood Alteration Anxiety/Agitation (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 7
Mood Alteration Depression (Nervous system disorders) | 3
Neuropathy Sensor (Nervous system disorders) | 19
Ocular Other (Eye disorders) | 1
Dry Eye (Eye disorders) | 2
Vision Flashing Lights/Floaters (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Abdominal Pain (General disorders) | 7
Pain Other (General disorders) | 4
Pain Tumor (General disorders) | 1
Headache (General disorders) | 6
Pelvic Pain (General disorders) | 1
Chest Pain (General disorders) | 2
Bone Pain (General disorders) | 2
Arthralgia (General disorders) | 4
Myalgia (General disorders) | 2
Pain Rectal/Perirectal (General disorders) | 1
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Urinary Frequency/Urgency (Renal and urinary disorders) | 2
Creatinine (Renal and urinary disorders) | 4
Renal/Gu Other (Renal and urinary disorders) | 2
Vaginitis No Infection (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Ureteral Obstruction (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less